CLINICAL TRIAL: NCT00996749
Title: Pilot Study to Determine the Optimal Dosage of Omega-3 Polyunsaturated Fatty Acid (PUFA) in Men With Advanced Prostate Cancer
Brief Title: Omega-3 Fatty Acids in Treating Patients With Advanced Prostate Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No Participants enrolled; slow accrual
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00014553; NCI-2009-01340 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 85108 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Stage III Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Fatty Acids, Omega-3; Fish Oils; Absorptiometry, Photon; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (omega-3 fatty acid) (Experimental): Patients receive long-term omega-3 PUFA supplementation PO.
  Interventions: Dietary Supplement: omega-3 fatty acid; Other: bone scan; Other: dual x-ray absorptometry; Other: laboratory biomarker analysis; Procedure: biopsy

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acid — Given PO
  Other Names: fish oil; n-3 fatty acid; O3FA
Other: bone scan — Correlative studies
Other: dual x-ray absorptometry — Correlative studies
  Other Names: DEXA scan; dual energy x-ray absorptometry
Other: laboratory biomarker analysis — Correlative studies
Procedure: biopsy — Correlative studies
  Other Names: biopsies

SUMMARY:
This phase I trial is studying the best way to give omega-3 fatty acids in treating patients with advanced prostate cancer. Omega-3 fatty acids may slow disease progression and may be an effective treatment for patients with advanced prostate cancer

DETAILED DESCRIPTION:
OBJECTIVES:

I. To conduct a pilot study of omega-3 polyunsaturated fatty acid (PUFA) (omega-3 fatty acid) supplementation in a group of patients with advanced prostate cancer to assess the dose of omega-3 PUFA necessary to achieve an omega-6 to -3 ratio of 1:1 on an individual basis and to assess the clinical impact of omega-3 supplementation on disease progression

OUTLINE:

Patients receive long-term omega-3 polyunsaturated fatty acid (PUFA) supplementation orally (PO).

After completion of study treatment, patients are followed up at 1, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

Disease is currently controlled with androgen ablation therapy Androgen ablation is expected to continue for at least 1 year Has been treated with androgen ablation therapy for at least 1 month Stable or decreasing prostate-specific antigen (PSA) on androgen ablation therapy Stable or no visible metastatic disease on imaging Eastern Cooperative Oncology Group (ECOG) functional status of at 0 or 1

Exclusion Criteria:

Eligible for local intervention with surgery or radiation Increasing serum PSA on hormonal ablation Radiographic evidence of progression of disease on hormonal ablation Current or history of second malignancy Previously treated with chemotherapeutic agents Previous history of intermittent androgen therapy Gastrointestinal (GI) disease that impacts absorption of nutrients

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Omega-3 fatty acid levels in serum and fat biopsies | At 1 year
Omega-6 fatty acid levels in serum and fat biopsies | At 1 year
Tolerability of omega-3 fatty acid supplementation | At 1 month
Tolerability of omega-3 fatty acid supplementation | At 6 months
Tolerability of omega-3 fatty acid supplementation | At 12 months

SECONDARY OUTCOMES:
Time to PSA progression | At 1 year
Rates of PSA progression | At 1 year
Status of bony metastasis | At baseline
Bone density as assessed by dual energy x-ray absorptiometry (DEXA) scan | At baseline
Bone density as assessed by DEXA scan | At 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Majid Mirzazadeh, Principal Investigator — Wake Forest University Health Sciences